CLINICAL TRIAL: NCT02683993
Title: Utilizing Holmium Laser for FURS Renal Stone Lithotripsy Comparing Stone Breaking vs. Stone Dusting Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUM-SBU-VP-15-01
Record Dates: First submitted 2016-01-28; First posted 2016-02-17 (Estimated); Results first posted 2025-11-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Stone Clearance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stone breaking (Experimental): Lithotripsy will be performed using the Lumenis Pulse 120H holmium laser system with low frequency parameters.
  Interventions: Device: Lumenis Pulse 120H holmium laser system and 200 DFL ball tip fiber
- Stone dusting (Experimental): Lithotripsy will be performed using the Lumenis Pulse 120H holmium laser system with high frequency parameters.
  Interventions: Device: Lumenis Pulse 120H holmium laser system and 200 DFL ball tip fiber

INTERVENTIONS:
Device: Lumenis Pulse 120H holmium laser system and 200 DFL ball tip fiber — The Lumenis Pulse P120H will be utilized in high and low frequencies according to subjects group allocation.

SUMMARY:
Twenty (20) subjects presenting with a renal stone and candidates for FURS (flexible ureteroscopic renal surgery) will undergo a single FURS procedure for a kidney stone as part of the study, using the study device. These subjects will be randomized into stone breaking treatment or stone dusting.

DETAILED DESCRIPTION:
This is a randomized, two-arm, prospective, single center study. Subjects will undergo a single flexible ureteroscopic renal surgery (FURS) procedure for a kidney stone as part of this study, using the study device, and will be treated as randomized to either stone breaking treatment or stone dusting treatment. Follow up visits are scheduled for the day of release from the hospital and at 1 month post procedure. Additional treatment sessions, if required, will be at the discretion of the investigator, as part of the site standard of practice. Additional treatment sessions will not be included in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject will be older than 18 years of age
2. Subject was diagnosed with renal calculi meeting the following criteria:

   * Largest stone measures no more than 2cm on a single diameter and is no less than 0.8cm as defined by X-ray or CT.
   * Accumulative stone burden (addition of all stone diameters) is no more than 2.5cm.
3. Subject is a candidate for FURS procedure
4. Subject is willing and has signed the Informed Consent Form

Exclusion Criteria:

1. Subject has undergone a previous treatment for stones in the same kidney
2. Subject requires another, concomitant procedure, other than FURS, to be performed during this treatment session.
3. Female subject is pregnant
4. Concomitant anticoagulant medication that cannot be suspended during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Miller, Study Director — Boston Scientific Corporation
Locations (1):
- New York Methodist Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stone Breaking | Stone Dusting
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stone Breaking | Stone Dusting | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (11.2) | 60.9 (15.4) | 61.6 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 8 | 5 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Stone Clearance
Description: stone clearance will be confirmed by CT or X-Ray at 1 month follow up.
Time Frame: Stone clearance based on 1 month follow-up imaging data
Measure: Count of Participants; unit: Participants
Arm/Group | Stone Breaking | Stone Dusting
Number analyzed (Participants) | 10 | 10
Participants
  Complete clearance | 6 | 6
  Evidence of fragments not requiring intervention | 3 | 4
  Evidence of fragments requiring an additional intervention | 1 | 0

2. Primary Outcome: Post-procedure Catheterization
Description: Post-procedure catheterization by group
Time Frame: Post-procedure through hospital discharge; typically discharge occurs on the same day or 1 day post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Stone Breaking | Stone Dusting
Number analyzed (Participants) | 10 | 10
Participants
  Ureteric catheter not placed at the end of procedure | 9 | 9
  Ureteric catheter placed at the end of procedure and not removed at hospital discharge | 1 | 0
  Ureteric catheter placed at the end of procedure; removal at hospital discharge unknown | 0 | 1

3. Primary Outcome: Procedure Time
Description: Duration (in minutes) of the procedure as an indicator for treatment efficiency.
Time Frame: during the procedure
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Stone Breaking | Stone Dusting
Number analyzed (Participants) | 10 | 10
Minutes | 46.3 (24.8) | 36.1 (16.5)

4. Primary Outcome: Usage of Alternative Stone Extracting Devices
Description: The need of the surgeon to use baskets, forceps or saline flushing to achieve complete stone clearance. This outcome can influence both procedure time and further complication.
Time Frame: as measured during the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Stone Breaking | Stone Dusting
Number analyzed (Participants) | 10 | 10
Participants
  Any alternate stone extracting devices used | 0 | 1
  No alternate stone extracting devices used | 10 | 9

5. Primary Outcome: Hospital Stay
Description: Hospital duration was measured to evaluate treatment efficiency
Time Frame: Procedure through hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Stone Breaking | Stone Dusting
Number analyzed (Participants) | 10 | 10
Participants
  Same day hospital discharge | 10 | 8
  Next day hospital discharge | 0 | 2

6. Secondary Outcome: Number of Participants With Intraoperative Complications
Description: Number of participants with complications that occur during the procedure.
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Stone Breaking | Stone Dusting
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

7. Secondary Outcome: Visibility During Procedure
Description: Visibility during procedure by group, rating categories: Poor, Fair, Good, Very Good or Excellent
Time Frame: Intraprocedural
Measure: Count of Participants; unit: Participants
Arm/Group | Stone Breaking | Stone Dusting
Number analyzed (Participants) | 10 | 10
Participants
  Poor | 0 | 0
  Fair | 0 | 0
  Good | 0 | 1
  Very Good | 7 | 6
  Excellent | 3 | 3

8. Secondary Outcome: Number of Participants With Occurrence of Retropulsion
Description: Occurrence of retropulsion by group
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Stone Breaking | Stone Dusting
Number analyzed (Participants) | 10 | 10
Participants
  Did not occur | 8 | 10
  Occurred several times but could be controlled | 2 | 0
  Occurred several times and was difficult to control | 0 | 0
  Stone lost to retropulsion | 0 | 0

9. Secondary Outcome: Ability to Reach Stone Fragments
Description: Performance rating of ability to reach stone fragments by group
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Stone Breaking | Stone Dusting
Number analyzed (Participants) | 10 | 10
Participants
  Easily performed | 6 | 9
  Performed well | 4 | 1
  Performed with difficulty | 0 | 0
  Impossible to perform | 0 | 0

10. Secondary Outcome: Damage to Scope or Fiber
Description: Damage to scope or fiber by group
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Stone Breaking | Stone Dusting
Number analyzed (Participants) | 10 | 10
Participants
  Scope damage: Yes | 0 | 0
  Scope damage: No | 10 | 10
  Fiber damage: Yes | 0 | 0
  Fiber damage: No | 10 | 10

11. Secondary Outcome: Fiber Transmission
Description: Fiber transmission (preserving energy transmission during lasing) by group
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Stone Breaking | Stone Dusting
Number analyzed (Participants) | 10 | 10
Participants
  Easily performed | 8 | 9
  Performed well | 2 | 1
  Performed with difficulty | 0 | 0
  Impossible to perform | 0 | 0

ADVERSE EVENTS:
Time Frame: Intra-operative to 1 month post-procedure
Description: Adverse event information was collected via assessments at follow-up visits.
Arm/Group | Stone Breaking | Stone Dusting
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stone Breaking (N=10) | Stone Dusting (N=10)
Bleeding (Renal and urinary disorders) | 0 (0) | 1 (1) — Occasional hematuria
Other (General disorders) | 0 (0) | 1 (1) — minimal discomfort

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT02683993/Prot_SAP_000.pdf